CLINICAL TRIAL: NCT06997497
Title: A Phase 3, Randomized, Open-label, Multicenter Clinical Study to Evaluate the Safety and Efficacy of MK-1084, Cetuximab, and mFOLFOX6 Versus mFOLFOX6 With or Without Bevacizumab as First-line Treatment of Participants With KRAS G12C-mutant, Locally Advanced Unresectable or Metastatic Colorectal Cancer (KANDLELIT-012)
Brief Title: A Clinical Study of Calderasib (MK-1084) With Targeted Therapy and Chemotherapy in People With Colorectal Cancer (MK-1084-012/KANDLELIT-012)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1084-012; MK-1084-012 (Other: MSD); KANDLELIT-012 (Other: MSD); 2024-517232-22-00 (Registry Identifier: EU CT); U1111-1311-8311 (Registry Identifier: UTN); jRCT2031250265 (Registry Identifier: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Colon Adenocarcinoma; Rectal Adenocarcinoma
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Oxaliplatin; Leucovorin; Fluorouracil; Cetuximab; Bevacizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Calderasib + Cetuximab + mFOLFOX6 (Experimental): Participants will receive calderasib orally, cetuximab per label every 2 weeks (Q2W), and mFOLFOX6 chemotherapy: oxaliplatin per label every 2 weeks (Q2W), leucovorin or levofolinate calcium per label Q2W, and 5-fluorouracil (5-FU) per label Q2W. Treatment will continue until criteria for discontinuation is met.
  Interventions: Drug: Calderasib; Drug: Oxaliplatin; Drug: Leucovorin/levofolinate calcium; Drug: 5-Fluorouracil; Biological: Cetuximab
- mFOLFOX6 (Active Comparator): Participants will receive mFOLFOX6 chemotherapy: oxaliplatin per label Q2W, leucovorin or levofolinate calcium per label Q2W, and 5-fluorouracil (5-FU) per label Q2W. Participants may also receive bevacizumab or bevacizumab biosimilar Q2W at the investigator's discretion. Treatment will continue until criteria for discontinuation is met.
  Interventions: Drug: Oxaliplatin; Drug: Leucovorin/levofolinate calcium; Drug: 5-Fluorouracil; Drug: Bevacizumab; Drug: Bevacizumab biosimilar

INTERVENTIONS:
Drug: Calderasib — Oral tablet
  Other Names: MK-1084
  Arms: Calderasib + Cetuximab + mFOLFOX6
Drug: Oxaliplatin — Per label
Drug: Leucovorin/levofolinate calcium — Per label
Drug: 5-Fluorouracil — Per label
Biological: Cetuximab — Per label
  Other Names: Erbitux
  Arms: Calderasib + Cetuximab + mFOLFOX6
Drug: Bevacizumab — Per label
  Other Names: Avastin
  Arms: mFOLFOX6
Drug: Bevacizumab biosimilar — Per label
  Other Names: MVASI
  Arms: mFOLFOX6

SUMMARY:
Researchers are looking for other ways to treat locally advanced or metastatic colorectal cancer (mCRC) that is unresectable and has a gene mutation called KRAS G12C.

Standard (or usual) treatments for this type of colorectal cancer may include mFOLFOX6 with or without bevacizumab. Researchers want to learn if adding calderasib (the study medicine) and cetuximab to mFOLFOX6 can treat locally advanced or mCRC with the KRAS G12C mutation. Calderasib and cetuximab are targeted therapies.

The goals of this study are to learn:

* About the safety of calderasib with cetuximab and mFOLFOX6 and if people tolerate the treatments
* If people who receive calderasib with cetuximab and mFOLFOX6 live longer without mCRC growing or spreading compared to people who receive mFOLFOX6 with or without bevacizumab.

DETAILED DESCRIPTION:
This study will have 2 parts.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has a histologically confirmed diagnosis of locally advanced unresectable or metastatic (unresectable Stage III or Stage IV as defined by American Joint Committee on Cancer [AJCC] eighth edition) colorectal adenocarcinoma
* Part 2 only: Has not received systemic anticancer therapy for locally advanced unresectable or metastatic colorectal cancer
* Tumor tissue demonstrates presence of a Kirsten rat sarcoma viral oncogene homolog G12C (KRAS G12C) mutation
* Human immunodeficiency virus (HIV)-infected participants must have well controlled HIV on antiretroviral therapy (ART)
* Participants who are Hepatitis B surface antigen (HBsAg) positive are eligible if they have received hepatitis B virus (HBV) antiviral therapy and have undetectable HBV viral load
* Participants with history of hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has active inflammatory bowel disease requiring immunosuppressive medication or previous clear history of inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis, chronic diarrhea)
* Has uncontrolled, significant cardiovascular disease or cerebrovascular disease
* Has known dihydropyrimidine dehydrogenase (DPD) deficiency
* HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Has received prior systemic anticancer therapy including investigational agents within 4 weeks before randomization
* Has 1 or more conditions that, in the opinion of the investigator, make the participant ineligible for treatment with bevacizumab
* Has known additional malignancy that is progressing or has required active treatment within the past 3 years
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis or leptomeningeal disease
* Has active infection requiring systemic therapy
* Has not adequately recovered from major surgery or have ongoing surgical complications
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 477 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2029-03-28 (Estimated); Study Completion 2030-10-27 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Dose-Limiting Toxicity (DLT) | Up to approximately 28 days
  A DLT is defined as the occurrence of protocol-specified toxicities if assessed by the investigator to be possibly, probably, or definitely related to study intervention administration.
Part 1: Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 44 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Part 1: Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 44 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Progression Free Survival (PFS) | Up to approximately 44 months
  PFS is defined as the time from randomization to the first documented disease progression or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 3 years
  ORR is defined as a confirmed complete response (CR: the disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 as assessed by blinded independent central review (BICR). The percentage of participants who experience CR or PR as assessed by BICR will be presented.
Overall Survival (OS) | Up to approximately 5 years
  OS is defined as the time from randomization to death due to any cause.
Duration of Response (DOR) | Up to approximately 4 years
  For participants who demonstrate a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by BICR will be presented.
Part 2: Number of Participants with an Adverse Event (AE) | Up to approximately 5 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Part 2: Number of Participants who Discontinue Study Treatment Due to an AE | Up to approximately 5 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Change from Baseline in the European Organization for Research and Treatment of Cancer (EORTC)-Quality of Life Questionnaire-Core 30 (QLQ-C30) Global Health Status (Item 29) and Quality of Life (Item 30) Combined Score | Baseline and up to approximately 5 years
  The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to the questions regarding Global Health Status (GHS; "How would you rate your overall health during the past week?") and Quality of Life (QoL; "How would you rate your overall quality of life during the past week?") are scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The change from baseline in GHS (EORTC QLQ-C30 Item 29) and QoL (EORTC QLQ-C30 Item 30) combined score will be presented. A higher score indicates a better outcome.
Change from Baseline in the EORTC-QLQ-C30 Physical Functioning (Items 1-5) Combined Score | Baseline and up to approximately 5 years
  The EORTC QLQ-C30 is a cancer specific health-related quality-of-life questionnaire. Participant responses to 5 questions about their physical functioning (Items 1-5) are scored on a 4-point scale (1=Not at All to 4=Very Much). Higher scores indicate better physical functioning. The change from baseline in EORTC QLQ-C30 Physical Functioning (Items 1-5) combined score will be presented.
Change from Baseline in the EORTC-QLQ-C30 Role Functioning (Items 6 and 7) Combined Score | Baseline and up to approximately 5 years
  The EORTC QLQ-C30 is a cancer specific health-related quality-of-life questionnaire. The role functioning score is based on participant responses to questions scored on a 4-point scale (1=Not at All to 4=Very Much). Higher scores indicate better role functioning. The change from baseline in EORTC QLQ-C30 Role Functioning (Items 6 and 7) combined score will be presented.
Change from Baseline in the EORTC-QLQ-C30 Appetite Loss (Item 13) Score | Baseline and up to approximately 5 years
  The EORTC QLQ-C30 is a cancer specific health-related quality-of life questionnaire, including a single-item scale score for appetite loss (QLQ-C30 Item 13). For this item, individual responses to the question "Have you lacked appetite?" are given on a 4-point scale (1=Not at all; 4=Very much). Scores are transformed to a range from 0-100, with a lower score indicating a better outcome. The change from baseline in the EORTC QLQ-C30 appetite loss (Item 13) scale score will be presented.
Change from Baseline in the EORTC-Quality of Life Questionnaire-Colorectal Cancer-Specific 29 Items (QLQ-CR29) Bloating (Item 37) Score | Baseline and up to approximately 5 years
  The EORTC QLQ-CR29 is a health-related quality-of life questionnaire specific for colorectal cancer, including a single-item scale score for bloating (QLQ-CR29 Item 37). For this item, individual responses to the question "Did you have a bloated feeling in your abdomen?" are given on a 4-point scale (1=Not at all; 4=Very much). Scores are transformed to a range from 0-100, with a lower score indicating a better outcome. The change from baseline in the EORTC QLQ-CR29 bloating (Item 37) scale score will be presented.
Time to First Deterioration (TTD) in EORTC QLQ-C30 Global Health Status (Item 29) and Quality of Life (Item 30) Combined Score | Baseline and up to approximately 5 years
  The EORTC QLQ-C30 is a cancer specific health-related quality-of-life questionnaire. TTD is defined as the time from baseline to the first onset of a ≥10-point deterioration (decrease) from baseline in global health status (GHS) (EORTC QLQ-C30 Item 29) & quality of life (QoL) combined score (EORTC QLQ-C30 Item 30). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10-point negative change (decrease) from baseline in GHS and QoL combined score, will be presented. A longer TTD indicates a better outcome.
TTD in EORTC QLQ-C30 Physical Functioning (Items 1-5) Score | Baseline and up to approximately 5 years
  The EORTC QLQ-C30 is a cancer specific health-related quality-of-life questionnaire. TTD is defined as the time from baseline to the first onset of a ≥10-point deterioration (decrease) from baseline in physical functioning score (EORTC QLQ-C30 Items 1-5). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10-point negative change (decrease) from baseline in GHS and QoL combined score, will be presented. A longer TTD indicates a better outcome.
TTD in EORTC QLQ-C30 Role Functioning (Items 6 and 7) Score | Baseline and up to approximately 5 years
  The EORTC QLQ-C30 is a cancer specific health-related quality-of-life questionnaire. The role functioning score is based on participant responses to questions scored on a 4-point scale (1 = 'Not at All' to 4 = 'Very Much'). Higher scores indicate better role functioning. The TTD, as assessed based on a ≥10-point negative change (decrease) from baseline in role functioning score, will be presented. A longer TTD indicates a better outcome.
TTD in EORTC QLQ-C30 Appetite Loss (Item 13) Score | Baseline and up to approximately 5 years
  The EORTC QLQ-C30 is a cancer specific health-related quality-of-life questionnaire. TTD is defined as the time from baseline to the first onset of a ≥10-point deterioration (decrease) from baseline in appetite loss score (EORTC QLQ-C30 Item 13). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10-point negative change (decrease) from baseline in physical functioning score, will be presented. A longer TTD indicates a better outcome.
TTD in EORTC QLQ-CR29 Bloating (Item 37) Score | Baseline and up to approximately 5 years
  The EORTC QLQ-CR29 is a health-related quality-of life questionnaire specific for colorectal cancer, including a single-item scale score for bloating (QLQ-CR29 Item 37). TTD is defined as the time from baseline to the first onset of a ≥10-point deterioration (decrease) from baseline in bloating score (QLQ-CR29 Item 37). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10-point negative change (decrease) from baseline in appetite loss score, will be presented. A longer TTD indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (83):
- United States (5):
  - Orlando Health Cancer Institute ( Site 0065), Orlando, Florida
  - Norton Cancer Institute, Audubon Hospital Campus ( Site 0054), Louisville, Kentucky
  - Renown Regional Medical Center ( Site 0056), Reno, Nevada
  - John Theurer Cancer Center at Hackensack University Medical Center ( Site 0060), Hackensack, New Jersey
  - Miami Valley Hospital South ( Site 0075), Centerville, Ohio
- Argentina (4):
  - Hospital Italiano de Buenos Aires ( Site 0102), Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Instituto Alexander Fleming ( Site 0101), Mar del Plata, Buenos Aires
  - Fundacion Estudios Clinicos ( Site 0105), Rosario, Santa Fe Province
  - Hospital Privado Universitario de Córdoba ( Site 0108), Córdoba
- Australia (2):
  - Sunshine Coast University Hospital ( Site 0451), Birtinya, Queensland
  - Monash Health ( Site 0454), Clayton, Victoria
- Brazil (7):
  - Hospital de Câncer de Recife ( Site 0158), Recife, Pernambuco
  - Hospital de Caridade de Ijuí ( Site 0150), Ijuí, Rio Grande do Sul
  - Associação Hospitalar Beneficente São Vicente de Paulo ( Site 0153), Passo Fundo, Rio Grande do Sul
  - CEPEN - Centro de Pesquisa e Ensino em Oncologia de Santa Catarina ( Site 0157), Florianópolis, Santa Catarina
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto ( Site 0159), São José do Rio Preto, São Paulo
  - Instituto do Cancer Arnaldo Vieira de Carvalho ( Site 0160), São Paulo
  - IBCC - Núcleo de Pesquisa e Ensino ( Site 0154), São Paulo
- Princess Margaret Cancer Centre ( Site 0001), Toronto, Ontario, Canada
- China (9):
  - Anhui Provincial Cancer Hospital ( Site 0803), Hefei, Anhui
  - The First Affiliated Hospital of Xiamen University ( Site 0806), Xiamen, Fujian
  - Sun Yat-Sen University Cancer Center ( Site 0800), Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital ( Site 0812), Guangzhou, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital ( Site 0804), Nanning, Guangxi
  - The Third Xiangya Hospital of Central South University ( Site 0834), Changsha, Hunan
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School ( Site 0825), Nanjing, Jiangsu
  - Jinan Central Hospital ( Site 0817), Jinan, Shandong
  - Sichuan Cancer hospital. ( Site 0831), Chengdu, Sichuan
- Colombia (3):
  - Hospital Universitario San Ignacio ( Site 0254), Bogota, Cundinamarca
  - IMAT S.A.S ( Site 0252), Montería, Departamento de Córdoba
  - Oncologos Del Occidente ( Site 0255), Pereira, Risaralda Department
- Finland (2):
  - Tampere University Hospital ( Site 1001), Tampere, Pirkanmaa
  - Helsinki University Hospital - Comprehensive Cancer Center (HYKS - Syöpäkeskus) ( Site 1000), Helsinki, Uusimaa
- Centre François Baclesse ( Site 1061), Caen, Calvados, France
- Katholisches Marienkrankenhaus gGmbH ( Site 1103), Hamburg, Germany
- Hong Kong (2):
  - Prince of Wales Hospital. ( Site 0500), Hong Kong
  - Queen Mary Hospital ( Site 0501), Hong Kong
- Israel (4):
  - Rambam Health Care Campus ( Site 1253), Haifa
  - Hadassah Medical Center ( Site 1252), Jerusalem
  - Rabin Medical Center ( Site 1251), Petah Tikva
  - Sheba Medical Center ( Site 1254), Ramat Gan
- National Cancer Center Hospital ( Site 0850), Chūō, Tokyo, Japan
- Netherlands (2):
  - Radboudumc ( Site 1354), Nijmegen, Gelderland
  - Amphia Ziekenhuis, locatie Breda Molengracht ( Site 1352), Breda, North Brabant
- Wielkopolskie Centrum Onkologii im. Marii Skłodowskiej-Curie ( Site 1457), Poznan, Greater Poland Voivodeship, Poland
- Romania (5):
  - Institutul Oncologic Cluj ( Site 1502), Cluj-Napoca, Cluj
  - SC Radiotherapy Center Cluj SRL-Oncologie Medicala ( Site 1501), Cluj-Napoca, Cluj
  - Centrul de Oncologie Sfantul Nectarie-Medical ( Site 1500), Craiova, Dolj
  - Fundeni Clinical Institute-Medical Oncology ( Site 1504), Bucharest
  - Institutul Regional de Oncologie ( Site 1505), Iași
- National Cancer Centre Singapore ( Site 0650), Singapore, Central Singapore, Singapore
- South Korea (7):
  - National Cancer Center ( Site 0702), Goyang-si, Kyonggi-do
  - Seoul National University Bundang Hospital ( Site 0705), Seongnam-si, Kyonggi-do
  - The Catholic University of Korea St. Vincent s Hospital ( Site 0703), Suwon, Kyonggi-do
  - Samsung Medical Center ( Site 0708), Gangnam, Seoul
  - Asan Medical Center ( Site 0707), Songpa-gu, Seoul
  - Kyungpook National University Chilgok Hospital ( Site 0701), Buk-Gu, Taegu-Kwangyokshi
  - Seoul National University Hospital ( Site 0706), Seoul
- Spain (9):
  - Institut Català d'Oncologia (ICO) - Badalona ( Site 1552), Badalona, Barcelona
  - Hospital Universitario Marqués de Valdecilla ( Site 1551), Santander, Cantabria
  - Hospital Insular de Gran Canaria ( Site 1558), Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Central de Asturias ( Site 1550), Oviedo, Principality of Asturias
  - Hospital Universitari Vall d'Hebron ( Site 1553), Barcelona
  - HOSPITAL GENERAL UNIVERSITARIO GREGORIO MARAÑON ( Site 1554), Madrid
  - Hospital Clinico San Carlos ( Site 1555), Madrid
  - HOSPITAL UNIVERSITARIO VIRGEN DEL ROCIO ( Site 1556), Seville
  - Instituto Valenciano de Oncologia - IVO ( Site 1557), Valencia
- Taiwan (4):
  - National Cheng Kung University Hospital ( Site 0754), Tainan
  - National Taiwan University Hospital ( Site 0751), Taipei
  - Taipei Veterans General Hospital ( Site 0752), Taipei
  - Chang Gung Memorial Hospital - Linkou Branch ( Site 0753), Taoyuan District
- Ukraine (11):
  - MNE "Clinical Center of Oncology, Hematology, Transplantology and Palliative Care of CRC" ( Site 1706), Cherkasy, Cherkasy Oblast
  - RMNE "Bukovyna Clinical Oncology Center" ( Site 1709), Chernivtsi, Chernivetska Oblast
  - MNPE "Prykarpattia Clinical Oncology Center of Ivano-Frankivsk Regional Council" ( Site 1701), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - CNE "Regional Clinical Oncology Center of the Kirovohrad Regional Council" ( Site 1702), Kropyvnytskyi, Kirovohrad Oblast
  - MNPE LTMU Multidisc. Clin. Hosp. of Emerg. and Intens. Care ( Site 1708), Lviv, Lviv Oblast
  - MNE "Central City Hospital" ( Site 1711), Rivne, Rivne Oblast
  - ME "Volyn Regional Clinical Hospital" of the VRC ( Site 1712), Lutsk, Volyn Oblast
  - Uzhgorod Central City Clinical Hospital ( Site 1700), Uzhhorod, Zakarpattia Oblast
  - Medical Center "Universal Clinic "Oberig" of Limited Liability Company "Kapytal" ( Site 1704), Kyiv
  - SI "National Institute of Surgery and Transplantology named after O. O. Shalimov" ( Site 1713), Kyiv
  - LLC "MEDICAL CENTER DOBROBUT-CLINIC" ( Site 1703), Kyiv
- The Christie NHS Foundation Trust ( Site 1755), Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/